CLINICAL TRIAL: NCT03766945
Title: A Survey of Fatigue and QoL Among Gastric Cancer Patients Undergoing Major Abdominal Surgery
Brief Title: Fatigue and QoL Among Gastric Cancer Patients Undergoing Abdominal Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201705112RINB
Record Dates: First submitted 2018-11-22; First posted 2018-12-06 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-06

CONDITIONS: Gastric Cancer; Surgical Wound Infection; Fatigue; Quality of Life
Keywords: Gastric Cancer; Surgery; Fatigue; Quality of Life
MeSH Terms: conditions — Stomach Neoplasms; Surgical Wound Infection; Fatigue

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples Without DNA — Biomarkers including pre-operative and post-operative serum IFN-gamma, IL-1 beta, IL-4, IL-6, IL-10 and TNF.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: Cancer-related fatigue (CRF), one of the indicators of QoL, is one of the most common side effects of cancer and its treatment. However, the pathophysiological mechanisms involved in CRF among cancer patients are not completely understood. Therefore, more in-depth researches on CRF of surgical patients suffering from gastric cancer are needed in Taiwan.

Purpose: The purpose of this study is to examine the incidence rate and correlated factors (QoL and immune biomarkers) of CRF among gastric cancer patients undergoing major abdominal surgery.

Method: A longitudinal study was conducted to recruit gastric cancer patients who scheduled to operate at surgical clinics from a northern medical center in Taiwan. The data will be collected with a structured questionnaire and Immune markers assessments via purposive sampling of 120 subjects. Before operation, on day 1 after operation, and on day 7 after operation, the biomarkers will be measured. The BFI-T questionnaire will be filled out before surgery and on day 1, 2, 7, 28 after surgery; The EORTC QLQ-C30 and EORTC QLQ-STO22 questionnaire will be filled out before surgery and on day 7, 28 after surgery; Type D scale-14(Taiwanese version) questionnaire will be filled out before surgery and on day 28 after surgery. Data will be analyzed by using descriptive statistics, paired t-test, Chi square test, Pearson's correlation, and the generalized estimating equation (GEE) was used to identify significant factors with QoL after operation.

Anticipated achievement: The anticipated achievement of this study is to provide healthcare providers with more knowledge about CRF, and help them to enhance the quality of life on gastric cancer patients in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of gastric cancer and schedule for major abdominal surgery
2. Eastern Cooperative Oncology Group (ECOG) performance status ≤2

Exclusion Criteria:

1. Severe multiple organ impairment, comorbidities or immune disorder before surgery
2. Undergoing chemotherapy or radiotherapy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Gastric cancer patients who are scheduled for major abdominal surgery will be enrolled.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2017-07-27 (Actual); Primary Completion 2019-07-25 (Estimated); Study Completion 2019-07-25 (Estimated)

PRIMARY OUTCOMES:
Fatigue | Change from baseline fatigue at 1 month
  Brief Fatigue Inventory-Taiwan Form (BFI-T). The questionnaire includes 10 items to assess fatigue.

SECONDARY OUTCOMES:
Quality of Life | Change from baseline quality of life at 1 month
  Quality of Life Questionnaire(EORTC QLQ-C30 and EORTC QLQ-STO22 questionnaire). The questionnaire includes 52 items to assess quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Ming Wu, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No